CLINICAL TRIAL: NCT07373678
Title: Coronary Artery Bypass Surgery Versus Percutaneous Coronary Intervention in Patients With Isolated Chronic Total Occlusion of the Left Anterior Descending Artery: The RITUAL Study
Brief Title: CABG Versus PCI in Patients With Isolated LAD Chronic Total Occlusion
Acronym: RITUAL
Status: Completed | Type: Observational
Sponsor: Mersin Medicalpark Hastanesi (Other)
Collaborators: Biruni University (Other); Mersin Training and Research Hospital (Other Government); Necmettin Erbakan University (Other); Jolimont Hospital (Other); Minneapolis Heart Institute (Other)
Responsible Party: Principal Investigator, Sefa Sural, Assistant Professor of Cardiology, Mersin Medicalpark Hastanesi
Other Study IDs: MLP-SSURAL-002
Record Dates: First submitted 2026-01-17; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Total Occlusion
Keywords: Chronic total occlusion; Coronary artery bypass; Percutaneous coronary intervention; left anterior descending artery; isolated LAD CTO
MeSH Terms: interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Bypass Grafting (CABG): Patients with isolated chronic total occlusion of the left anterior descending artery who underwent coronary artery bypass graft surgery.
  Interventions: Procedure: Coronary Artery Bypass Grafting
- Percutaneous Coronary Intervention (PCI): Patients with isolated chronic total occlusion of the left anterior descending artery who underwent percutaneous coronary intervention.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — Coronary artery bypass graft surgery performed as part of routine clinical care prior to study inclusion.
  Groups: Coronary Artery Bypass Grafting (CABG)
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention performed as part of routine clinical care prior to study inclusion.
  Groups: Percutaneous Coronary Intervention (PCI)

SUMMARY:
The aim of this study is to compare coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI) in the treatment of isolated chronic total occlusion (CTO) of the left anterior descending (LAD) artery in terms of short- and mid-term clinical outcomes, myocardial revascularization success, and complication rates.

DETAILED DESCRIPTION:
Chronic total occlusion (CTO) represents one of the most challenging subgroups of coronary artery disease and is closely associated with adverse cardiovascular outcomes. Previous studies have demonstrated that patients with CTO experience a higher incidence of major adverse cardiovascular events compared with patients without CTO but with significant coronary artery disease (CAD), even after adjustment for demographic characteristics, clinical parameters, and disease severity. Among these patients, those with unrevascularized CTO constitute the highest-risk group, whereas successful revascularization has been shown to reduce the risk to a level comparable to that of patients without CTO but with significant CAD.

Among CTOs, isolated total occlusion of the left anterior descending (LAD) artery has particular clinical importance due to its critical role in myocardial perfusion. Two main revascularization strategies are currently used in the treatment of isolated LAD CTO: percutaneous coronary intervention (PCI) and single-vessel coronary artery bypass grafting (CABG). In surgical revascularization, the left internal mammary artery (LIMA) is most commonly used, although saphenous vein grafts may be preferred in selected cases.

However, direct comparative data between these two treatment strategies in this specific patient population remain extremely limited. In particular, differences between CTO-PCI and single-vessel CABG with respect to revascularization success, in-hospital events, and early post-discharge outcomes have not been systematically evaluated. In the present study, within the framework of the RITUAL study, the outcomes of CTO-PCI and CABG surgery were compared in patients with isolated LAD CTO.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of the index procedure.
* Diagnosis of isolated chronic total occlusion (CTO) of the left anterior descending (LAD) coronary artery.
* Isolated LAD CTO defined as a de novo or in-stent total occlusion confined to the LAD artery, without significant coronary artery disease (defined as ≥50% stenosis) in other major epicardial coronary arteries, including the left circumflex (LCx), right coronary artery (RCA), or major side branches.
* No prior percutaneous coronary intervention (PCI) performed in non-LAD coronary arteries.
* Patients who underwent coronary revascularization with either coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) for isolated LAD CTO.

Exclusion Criteria:

* History of malignancy or active malignant disease at the time of the index procedure.
* Prior coronary artery bypass grafting (CABG) or prior percutaneous coronary intervention (PCI) performed in non-LAD coronary arteries.
* Presentation with ST-segment elevation myocardial infarction (STEMI).
* Discontinuation of prescribed medical therapy by patient preference within one year after the index procedure.
* Presence of multiple chronic total occlusions (CTOs) involving more than one coronary artery.
* Significant side branch disease of the LAD requiring two bypass grafts.
* Performance of crossover stenting from the LAD into the left main coronary artery during LAD CTO-PCI.
* Treatment of LAD CTO with drug-eluting balloon (DEB) angioplasty without stent implantation.
* Left ventricular ejection fraction (LVEF) less than 30%.
* Presence of severe valvular heart disease (e.g., severe aortic or mitral stenosis or regurgitation).
* Incomplete angiographic or clinical follow-up data.
* Use of mechanical circulatory support devices due to advanced heart failure, including intra-aortic balloon pump (IABP), extracorporeal membrane oxygenation (ECMO), or left ventricular assist device (LVAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older with isolated chronic total occlusion (CTO) of the left anterior descending (LAD) coronary artery who underwent coronary revascularization with either coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) as part of routine clinical care. Isolated LAD CTO was defined as a de novo or in-stent total occlusion confined to the LAD artery, without significant coronary artery disease (≥50% stenosis) in other major epicardial coronary arteries. Patients with prior coronary revascularization, multiple CTOs, severe left ventricular dysfunction, or incomplete follow-up data were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Procedural success | perioperatively / periprocedurally
  Successful completion of coronary revascularization of the left anterior descending artery without in-hospital major adverse cardiac events.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACCE) at 3 years | 3 years
  Composite endpoint including all-cause mortality, non-fatal myocardial infarction, cerebrovascular events, and target vessel revascularization within 3 years after the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sefa SURAL, MD, Principal Investigator — Toros University
Locations (1):
- Sefa SURAL, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the retrospective design of the study and institutional data privacy policies.